CLINICAL TRIAL: NCT05519722
Title: The Effects of an Expectation-focused Nonguided Therapy Preparation
Acronym: ENThER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENThER
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Expectations
Keywords: expectations; intervention; online; psychotherapy; patients; waitlist

STUDY DESIGN:
Intervention Model Description: The patients will be randomly distributed to the intervention group or the control group. The intervention group will receive a nonguided online-intervention to optimize expectations. The control group will receive no intervention at all.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Expectation-focused online intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Expectation-focused online intervention — Patients receive an expectation-focused online intervention (around 30 minutes) consisting of a video with general information about psychotherapy, a video with reports of patients' therapy experiences, questions on the content of the videos as well as open questions on personal strengths, fears and expectations in the context of therapy. This intervention aims to optimize patients' expectations by focusing on positive and realistic expectations regarding the psychotherapeutic process.
  Arms: Intervention group

SUMMARY:
Various studies have shown that a more positive outcome expectation can have an influence on the actual treatment outcome of outpatient psychotherapeutic treatments. Therefore, the aim of this online study is to investigate whether [1] the patients' outcome expectation of outpatient psychotherapy can be optimized by a brief nonguided online intervention and whether [2] this intervention can influence important factors of psychotherapy, such as active cooperation, the therapeutic relationship, motivation, and regular attendance to therapy.

To examine these questions, patients who are waiting for outpatient therapy will be randomized into two groups (control vs. intervention group) after baseline assessment. The intervention group will participate in a brief therapy preparation (30 minutes) that focuses on optimizing outcome expectations. Both groups will fill out questionnaires again on the following day, during the diagnostic phase at the beginning of therapy and six months later (or at the end of therapy in case therapy ends before the 6-month-follow-up). Furthermore, therapists will also fill out questionnaires during the diagnostic phase at the beginning of therapy and six months later (or at the end of therapy in case therapy ends before the 6-month-follow-up).

ELIGIBILITY:
Inclusion Criteria:

* patients who are waiting for therapy at the ambulance for psychotherapy Marburg ("Psychotherapie-Ambulanz Marburg")
* Age 18 or above
* Fluency in German
* Informed consent

Exclusion Criteria:

* visual or hearing impairment that interferes with viewing or listening to video recordings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in outcome expectation (Credibility and Expectancy Questionnaire (CEQ) scale) from Baseline to T1 | Baseline, T1 (following day)
  German version of the Credibility and Expectancy Questionnaire (CEQ), 6-item scale (Raeke, 2013).The CEQ consists of two subscales with four items measuring cognitive-focused credibility (e.g., "At this point, how logical does the therapy offered to you seem?") and two items measuring affect-focused expectations (e.g., "By the end of the therapy period, how much improvement in your symptoms do you really feel will occur?"). The CEQ applies different rating scales; a 9-point scale ranging from 1 (not at all) to 9 (very much) and a percentage rating scale ranging from 0% (not at all) to 100% (very much) with higher sum scores indicating greater treatment credibility and expectations.

SECONDARY OUTCOMES:
Change in outcome expectation (Credibility and Expectancy Questionnaire (CEQ) scale) from Baseline to T2 to T3 | Baseline, T2 (start of therapy), T3 (6-month-follow-up)
  German version of the Credibility and Expectancy Questionnaire (CEQ), 6-item scale (Raeke, 2013).The CEQ consists of two subscales with four items measuring cognitive-focused credibility (e.g., "At this point, how logical does the therapy offered to you seem?") and two items measuring affect-focused expectations (e.g., "By the end of the therapy period, how much improvement in your symptoms do you really feel will occur?"). The CEQ applies different rating scales; a 9-point scale ranging from 1 (not at all) to 9 (very much) and a percentage rating scale ranging from 0% (not at all) to 100% (very much) with higher sum scores indicating greater treatment credibility and expectations.
Change in outcome expectation and process expectations (Milwaukee Psychotherapy Expectations Questionnaire (MPEQ)) from Baseline to T1 to T2 to T3 | Baseline, T1 (following day), T2 (start of therapy), T3 (6-month-follow-up)
  German version of the Milwaukee Psychotherapy Expectations Questionnaire (MPEQ), measures outcome expectations and process expectations (Norberg et al., 2011) with four outcome expectation questions, ask about expected improvements in self-respect, strength to avoid feelings of distress, being a better person, and being a more optimistic person by the end of therapy.
Change in scores on the subscale for treatment expectations of the the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) from baseline to T1 to T2 to T3 | Baseline, T1 (following day), T2 (start of therapy), T3 (6-month-follow-up)
  Prior experiences with psychotherapy and treatment expectations are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences and subscale for treatment expectations (Rief et al., 2021). Answers are provided on a numeric rating scale ranging from 0 to 10.
Change in symptom severity (Beck Depression Inventory (BDI-II), Patient Health Questionnaire 4 (PHQ-4), Symptom Checklist-90-Revised (SCL-90-R)) | Baseline, T2 (start of therapy), T3 (6-month-follow-up)
  BDI-II:
  Self-report questionnaire to assess subjective depression symptomatology; 21 items (each item response is scored 0-3); total scores range from 0 - 63 (higher scores indicate more depressiveness)
  SCL-90-R:
  Self-report questionnaire to evaluate a broad range of psychological problems and symptoms of psychopathology, 90 items, 5-point rating scale.
  PHQ-4:
  Self-report questionnaire to screen for psychological distress, 4-point rating scale, total scores range from 0 - 12, subscales for depression and anxiety range from 0 - 6.

OTHER OUTCOMES:
General Self-Efficacy Scale (GSE) | Baseline, T1 (following day), T2 (start of therapy), T3 (6-month-follow-up)
  Self-efficacy via the German version of the General Self-Efficacy Scale (GSE), a 10-item scale measuring general self-efficacy. 10 items, 4-point Likert-scale ranging from 1 to 4, total score ranges from 10 - 40 with high scores indicating high levels of general self efficacy perceptions.
Therapeutic Relationship (Helping Alliance Questionaire (HAQ)) | T2 (start of therapy), T3 (6-month-follow-up)
  HAQ is a self-report questionnaire made up from 12 questions concerning the perceived therapeutic relationship and the therapeutic process can be answered as well by the patient as by the therapist. 6-point rating scale, total score and two subscales ("relation to the therapist" and "satisfaction with therapeutic outcome").
Treatment adherence | T2 (start of therapy), T3 (6-month-follow-up)
  active participation in and between therapy sessions, count of missed sessions
Patients' Illness Perception (Brief Illness Perception Questionnaire, B-IPQ) | Baseline, T1 (following day), T2 (start of therapy), T3 (6-month-follow-up)
  The B-IPQ surveys the cognitive and emotional representations of illness. Item 1-5 measure cognitive illness representations (consequences, timeline, personal control, treatment control, and identity). Item 6 and 8 quantify emotional representations (concern & emotions). Item 7 assesses illness comprehensibility. Item 9 is an open question (three most important causal factors in their illness). Items range from 0-10.
Previous treatment experiences on the subscale for previous treatment experiences of the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) | Baseline
  Prior experiences with psychotherapy are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences (Rief et al., 2021). Answers are provided on a numeric rating scale ranging from 0 to 10.
Social Support (ESSI-D) | T1 (following day), T2 (start of therapy), T3 (6-month-follow-up)
  The german version of the 5-item version of the "ENRICHD Social Support Instrument" (ESSI) measures the perceived social support, 5-point Likert-scale.
Personality (Big Five Inventory, BFI-10) | Baseline
  Items range from 1 - 5. The questionnaire includes the scales "openness to experience", "conscientiousness", "extraversion", agreeableness and neuroticism.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Clinical Psychology and Psychotherapy Dept. of Psychology, Philipps-University Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data will be shared with researchers providing a relevant and methodologically sound proposal